CLINICAL TRIAL: NCT01348204
Title: Nasal Potential Studies Utilizing CFTR Modulators (UAB Center for Clinical and Translational Science)
Brief Title: Nasal Potential Studies Utilizing Cystic Fibrosis Transmembrane Regulator (CFTR) Modulators
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Dr. Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: F100107002
Record Dates: First submitted 2010-06-01; First posted 2011-05-05 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- quercetin (Experimental): health food supplement
  Interventions: Other: quercetin

INTERVENTIONS:
Other: quercetin — health food supplement

SUMMARY:
The purpose of the study is to develop new biomarkers for studies of cystic fibrosis (CF). Defects in the gene encoding Cystic Fibrosis Transmembrane Regulator (CFTR) cause CF, an autosomal recessive disorder affecting mainly the pulmonary and digestive tract, leading to early death largely due to progressive loss of pulmonary function. In vitro experiments show that quercetin - a dietary supplement with a well-established safety profile for human use, including clinical trials in a variety of disorders encompassing cancer, heart disease, and as an anti-inflammatory agent - induces activation of CFTR. The nasal potential difference (NPD) test is a measurement of voltage across the nasal membrane and as a fundamental biomarker for CFTR activity in vivo. The NPD is a useful, well-established tool in CF research to determine both diagnoses as well as to measure the effect of new therapies. In vitro experiments show that quercetin induces activation of CFTR additive to that seen with current NPD reagents. In addition, it activates rescued mutant CFTR in vitro (∆F508 CFTR the most common cause of CF), whereas conventional agonists do not. Preliminary in vivo experiments mirrored these results and show that quercetin activates CFTR in human (n=12) NPD tests. Importantly, quercetin perfusion was well-tolerated by a validated sinus questionnaire and physician assessed nasal examination rating. These studies provide strong support for use of quercetin as potentiator of CFTR Cl- channel function by nasal administration. By adding quercetin to the sequence of perfusion solutions for NPD, the investigators may be better suited to detect ∆F508 CFTR activity of rescued mutant protein in the CF patient population.

DETAILED DESCRIPTION:
Flavonoids are a large group of naturally occurring polyphenolic compounds which are ubiquitous throughout the plant kingdom and are bio-available in fruits, vegetables, nuts, seeds, flowers, and bark. Quercetin has raised particular interest as it is not only a major component of the naturally occurring dietary flavonols, but it also seems to have anti-oxidant, anti-carcinogenic, anti-inflammatory, as well as cardioprotective functions. Recently, our laboratory and others have reported that quercetin, in addition to its other functions, plays a role in improving the function of chloride (Cl-) transport in the (CFTR).

It is well established that genistein, a flavone related to quercetin, increases mutant and wild-type CFTR channel activity. Genistein is now widely used in various cell systems, tissues, and species as a robust CFTR activator. Although it has been extremely helpful in laboratory experiments, Genistein translates poorly into human experiments as it has poor dissolution in solvent. As almost all flavonoids activate CFTR, deeper examination of other members of this family is important for both clinical use as well as a tool for future clinical studies. Quercetin is now available in health food stores as a dietary supplement in both pill as well as beverage form. It may also be beneficial for the treatment of CF and for use as a direct activator of CFTR for use in clinical trials where measurements of CFTR activity are important.

Through a better understanding of CFTR biogenesis and activation, new therapeutic approaches that restore activity to mutant CFTR molecules in vitro and in vivo are being developed. Biomarkers that can detect activity of rescued CFTR are required to measure therapeutic effects of new compounds. Current methods have yet to show consistent rescue of CFTR activity, raising the importance of optimizing detection strategies, including the most effective NPD endpoint. This may be particularly important for subjects harboring the ∆F508 mutation which in addition to its cell processing abnormality, also exhibits a channel gating defect (it does not activate with the conventional NPD agonist isoproterenol) thereby reducing detection of rescued protein. The investigators have previous experience evaluating alternative CFTR activating agents, both in CF animal models, and in human subjects. By adding quercetin to the sequence of perfusion solutions for NPD, the investigators may be better suited to detect CFTR activity of rescued mutant protein. In vitro experiments show that quercetin induces activation of CFTR additive to that seen with current NPD reagents. Preliminary in vivo experiments of non-CF individuals mirrored these results and show that quercetin activates CFTR in human NPD tests (n=12). Importantly, quercetin perfusion was well-tolerated by a validated sinus questionnaire and physician assessed nasal examination rating. As preliminary data suggest perfusion of quercetin may improve defective CFTR activation in surface localized ΔF508, use of this agent within an NPD protocol is likely to improve detection of ΔF508 CFTR resident at the cell surface, representing a potential means to identify new candidates for systemic CFTR potentiator therapies.

ELIGIBILITY:
Inclusion Criteria:

* 8-65 years old
* absence of pulmonary exacerbation in the last 2 weeks
* willingness to perform nasal potential difference measurement

Exclusion Criteria:

* Need for chronic oxygen supplementation
* positive for B. cepecia within the last year
* active participation in another interventional trial utilizing ion transport modulators
* interfering medical conditions
* pregnant females

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
NPD Biomarker | patients enroll for a single 2-4 hour visit
  Determine whether the NPD biomarker can be improved by including the potentiator quercetin to activate CFTR dependent ion channel activity among CF individuals with surface localized CFTR mutations

SECONDARY OUTCOMES:
Residual CFTR activity | patients enroll for a single 2-4 hour visit
  Determine the relationship between quercetin induced residual CFTR activity (detected in CF patients by the NPD biomarker) and stimulated short circuit currents (Isc) in primary airway cultures harvested from CF tissue donors.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Rowe, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States